CLINICAL TRIAL: NCT00407147
Title: ProBac - Use of Procalcitonin Level as Part of a Decision Tree to Discontinue Antibiotics When Started Empirically in the ICU in Hemodynamically Stable Patients With no Site of Infection Identified
Brief Title: Procalcitonin Level to Discontinue Antibiotics on ICU Patients With no Obvious Site of Infection
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: termination due to futility (very slow patient enrollment)
Sponsor: Brahms AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ProBac
Record Dates: First submitted 2006-11-29; First posted 2006-12-04 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Infection; Bacterial Infection; Sepsis
Keywords: bacterial infection; empiric antibiotic treatment; duration antibiotic treatment; reduce antibiotic treatment; procalcitonin; PCT Kryptor; sepsis; Intensive Care Unit; antibiotic treatment
MeSH Terms: conditions — Infections; Bacterial Infections; Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Standard treatment
- PCT (Experimental): PCT guided arm
  Interventions: Device: Procalcitonin assay - B.R.A.H.M.S PCT sensitive Kryptor

INTERVENTIONS:
Device: Procalcitonin assay - B.R.A.H.M.S PCT sensitive Kryptor — antibiotic treatment based on clinical decision making with "traditional thought processes" used in both groups. In addition the physician will be given access to Procalcitonin values with recommended thresholds for likelihood of infection.
  Other Names: B.R.A.H.M.S, Kryptor, Procalcitonin
  Arms: PCT

SUMMARY:
The purpose of this study is to test whether a U.S. Food and Drug Administration (FDA) approved laboratory test (PCT Kryptor) can help doctors make better decisions on the need for antibiotic therapy in ICU patients with suspected infections.

DETAILED DESCRIPTION:
The study is undertaken as prospective, randomized, controlled, multicenter trial. The study population, ICU patients with empiric antibiotic treatment due to suspected but unproven infection, is randomly assigned to either a Standard Care Group or a Procalcitonin (PCT) Guided Group. In the standard care group, antibiotic treatment would be based totally on clinical decision making with "traditional thought processes" (i.e., cultures, response to antibiotics, risk of untreated infection, other laboratory findings, etc.). The PCT guided group will use the same "traditional thought processes" and in addition the physician will be given access to a PCT value for Day 1 and Day 4 along with the recommended thresholds for likelihood of infection. In conjunction with other laboratory findings and clinical assessments the threshold of PCT is used to continue or discontinue empiric antibiotic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Suspected infection (no clear-cut source of infection) as defined by the treating physician
* Empiric antibiotic treatment
* No clear-cut source of infection by clinical or microbiological criteria
* ICU patient
* Informed consent

Exclusion Criteria:

* Age <18 years
* Pregnancy
* Hemodynamic instability defined as persistent hypotension, need for on-going aggressive resuscitation and/or vasopressor support to maintain an adequate mean arterial blood pressure
* Need for antibiotic prophylaxis
* Patient withdrawn from empiric antibiotic treatment before Day 4
* Severely immuno-compromised patient (liver cirrhosis (Child-Pugh class C), immunosuppressive drugs after transplantation, neutropenia (absolute neutrophil count <1000 counts/L), CD-4 count less than 200)
* Patient with suspected bacterial or fungal endocarditis
* Patient with suspected meningitis
* Cardiopulmonary bypass within the last 7 days1)
* Major surgery within the last 7 days (surgery that induces a major inflammatory response such as heart or aortic surgery or major abdominal surgery (i.e. duodenopancreatectomy) or any surgery requiring massive blood transfusion.)
* Multiple trauma within the last 7 days
* Cardiopulmonary resuscitation (CPR) within the last 7 days
* Burns >20% body surface area
* Patient in terminal status referred for palliative care
* Patient with advanced directives or Do Not Resuscitate (DNR) orders
* Patient who is already enrolled in another therapeutic clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Days on antibiotics beginning with day 4 until the first day without antibiotics (up to max. 28 days follow up) | 28 days

SECONDARY OUTCOMES:
Days on antibiotics during ICU stay | up to 28 days
Sepsis classification | up to 28 days
SOFA score (modified) | up to 28 days
ICU or hospital mortality up to 28 days | up to 28 days
Frequency of infections | up to 28 days
ICU and hospital length of stay | up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Phil Dellinger, M.D., Study Chair — The Cooper Health System
Locations (3):
- United States (3):
  - Saint Louis University - medical intensive care unit, St Louis, Missouri
  - Cooper University Hospital, Camden, New Jersey
  - Rhode Island Hospital, Providence, Rhode Island

REFERENCES:
- [Background] Vincent JL, Bihari DJ, Suter PM, Bruining HA, White J, Nicolas-Chanoin MH, Wolff M, Spencer RC, Hemmer M. The prevalence of nosocomial infection in intensive care units in Europe. Results of the European Prevalence of Infection in Intensive Care (EPIC) Study. EPIC International Advisory Committee. JAMA. 1995 Aug 23-30;274(8):639-44. PMID 7637145
- [Background] Garnacho-Montero J, Garcia-Garmendia JL, Barrero-Almodovar A, Jimenez-Jimenez FJ, Perez-Paredes C, Ortiz-Leyba C. Impact of adequate empirical antibiotic therapy on the outcome of patients admitted to the intensive care unit with sepsis. Crit Care Med. 2003 Dec;31(12):2742-51. doi: 10.1097/01.CCM.0000098031.24329.10. PMID 14668610
- [Background] Christ-Crain M, Jaccard-Stolz D, Bingisser R, Gencay MM, Huber PR, Tamm M, Muller B. Effect of procalcitonin-guided treatment on antibiotic use and outcome in lower respiratory tract infections: cluster-randomised, single-blinded intervention trial. Lancet. 2004 Feb 21;363(9409):600-7. doi: 10.1016/S0140-6736(04)15591-8. PMID 14987884
- [Background] Rau B, Steinbach G, Gansauge F, Mayer JM, Grunert A, Beger HG. The potential role of procalcitonin and interleukin 8 in the prediction of infected necrosis in acute pancreatitis. Gut. 1997 Dec;41(6):832-40. doi: 10.1136/gut.41.6.832. PMID 9462219
- [Background] Meisner M, Tschaikowsky K, Palmaers T, Schmidt J. Comparison of procalcitonin (PCT) and C-reactive protein (CRP) plasma concentrations at different SOFA scores during the course of sepsis and MODS. Crit Care. 1999;3(1):45-50. doi: 10.1186/cc306. PMID 11056723
- [Background] Bergmans DC, Bonten MJ, Gaillard CA, van Tiel FH, van der Geest S, de Leeuw PW, Stobberingh EE. Indications for antibiotic use in ICU patients: a one-year prospective surveillance. J Antimicrob Chemother. 1997 Apr;39(4):527-35. doi: 10.1093/jac/39.4.527. PMID 9145828
- [Background] Roder BL, Nielsen SL, Magnussen P, Engquist A, Frimodt-Moller N. Antibiotic usage in an intensive care unit in a Danish university hospital. J Antimicrob Chemother. 1993 Oct;32(4):633-42. doi: 10.1093/jac/32.4.633. PMID 8288506
- [Background] Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Crit Care Med. 1985 Oct;13(10):818-29. PMID 3928249